CLINICAL TRIAL: NCT05772000
Title: Clinical Significance of Occult Central Nervous System Localization in Adult Patients With Acute Lymphoblastic Leukemia. Prospective, Multicenter Study.
Brief Title: Clinical Significance of Occult Central Nervous System Localization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Maria Ilaria Del Principe, Associate Professor, University of Rome Tor Vergata
Other Study IDs: CampusALL2022
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cerebrospinal fluids exams — cerebrospinal fluids will be examined by conventional cytology and flow cytometry

SUMMARY:
In acute lymphoblastic leukemia (ALL), the occult central nervous system (CNS) involvement appears to be associated with poor prognosis. Flow cytometry (FCM) allows detection of occult CNS localization. The current international guidelines do not recommend the use of FCM in the assessment of CNS at onset in adult ALL patients. Large-scale prospective studies will help to clarify whether or not patients with occult CNS localization should undergo CNS-directed therapy. Understanding this seems particularly important nowadays considering that with the introduction of new drugs (monoclonal antibodies, next-generation tyrosine kinase inhibitors, CAR-T) the therapeutic approach of patients with ALS is increasingly "chemo-free"

DETAILED DESCRIPTION:
The investigators propose a multicenter prospective study to evaluate the incidence of occult CNS localization and the impact of such localization on clinical outcome.Adult ALL patients routinely undergo diagnostic lumbar puncture (PL); cerebrospinal fluids (CSF )samples will be studied by investigation of conventional cytology (CC) and FCM at the time of the first and subsequent diagnostic PLs.

ELIGIBILITY:
Inclusion criteria.

* Patients aged more than18 years with diagnosis of ALL at onset undergoing diagnostic-therapeutic PL.
* Signed written informed consent in accordance with ICH/EU/GCP guidelines and national and local laws.

Exclusion criteria.

* Patients <18 years of age
* Diagnosis other than ALL
* Inability to perform PL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients affected by acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2024-09-08 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of occult CNS localization in adult patients with ALL | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ilaria Del Principe, Prof, Principal Investigator — University of Rome Tor Vergata
Locations (1):
- Tor Vergata University, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05772000/Prot_SAP_001.pdf